CLINICAL TRIAL: NCT01414842
Title: Randomized Controlled Study on the Effect of the Hemodiafiltration Plasma Sodium Biofeedback System on Cardiovascular Stability in Hemodialysis Patients
Brief Title: HFR A-equilibrium on Cardiovascular Stability
Acronym: AIMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera di Lecco (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Centre Pasteur Vallery Radot (Unknown)
Responsible Party: Principal Investigator, Francesco Locatelli, Prof., Azienda Ospedaliera di Lecco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HFR-AE-2006; HFR-BFBCK0611 (Other: AOLecco)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2007-01

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Standard constant (no profiled) sodium dialysate used during endogenous hemodiafiltration
  Interventions: Device: Standard sodium dialysate
- Automated profiled (Experimental): Automate sodium profiling in endogenous hemodiafiltration
  Interventions: Device: Automated sodium profiling in endogenous hemodiafiltration

INTERVENTIONS:
Device: Automated sodium profiling in endogenous hemodiafiltration — Automated sodium profiling during endogenous reinfusion hemodiafiltration technique. The device processes the dialysate sodium and ultrafiltration rate during dialysis to achieve a preset sodium target at the end of the treatment. Sodium dialysate and maximal ultrafiltration rate are constraint within safety limits during dialysis.
  Other Names: HFR-Aequilibrium
  Arms: Automated profiled
Device: Standard sodium dialysate — Standard constant (no profiled) sodium dialysate used during endogenous hemodiafiltration
  Other Names: Standard HFR
  Arms: Standard

SUMMARY:
Aim of the present randomized controlled multinational trial is the comparison of a novel biofeedback system on sodium profiling applied to a endogenous hemodiafiltration therapy, with the standard (no sodium profiling) hemodiafiltration technique on the intradialytic overall and cardiovascular stability.

DETAILED DESCRIPTION:
Online hemodiafiltration (OL-HDF) has been recently associated with better patient survival in comparison with standard hemodialysis in some large observational studies (Canaud et al, KI, 2006; Vilar et al, CJASN , 2009) supporting the hypothesis that convection can improve patients outcomes. Moreover, it has been demonstrated in randomized controlled trials (Locatelli et al, Journal American Society of Nephrology, 2010) that OL-HDF significantly reduced the frequency of intradialytic hypotension. Nonetheless, the associated comorbidities and ageing of dialysis population require further devices able to improve treatment tolerance. Among these tools, the sodium profiling and biofeedback system seem to be promising to accomplish this task. But the correct intradialytic sodium balance is still far away today to be easily achieved. The use of an automated adaptive system dialysis to the sodium profiling has been investigated in a feasibility trial (Colì et al International Journal Artificial Organs, 2003). They also investigated the impact of such a device on treatment tolerance.

The aim of this randomized multinational multicenter controlled trial is to evaluate the impact of sodium profiling applied to a endogenous hemodiafiltration technique on the intradialytic cardiovascular stability in comparison to standard no profiled endogenous hemodiafiltration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 30% of dialysis complicated by hypotension
* age between 18 and 85 yers
* time on dialysis greater than 6 months
* residual creatinine clearance less than 2 ml/min/1.73 m2
* native fistula or central venous catheter with blood flow rate greater than 250 ml/min

Exclusion Criteria:

* Life expectancy less than 1 year
* solid active neoplasm
* pregnancy
* major event in the previous 3 months (ictus, myocardial infarction, cachexia)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of dialysis complicated by at least one hypotension | six months
  Hypotension definition:
  If predialysis systolic blood pressure greater than100 mmHg then a value during dialysis below 90 mmHg or any systolic blood pressure reduction greater than 25 mmHg in presence of symptoms or If predialysis systolic blood pressure less than 90 mmHg a reduction of at least 10% accompanied by symptoms

SECONDARY OUTCOMES:
Blood Pressure Intradialytic symptoms | six months
  Systolic, diastolic blood pressures (SBP, DBP) and heart rate (HR) measured at the beginning of each treatment and every 30 minutes till the end of dialysis; intradialytic symptoms (nausea, vomiting, hypotension, headache, cramps) and related clinical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Locatelli, Prof., Study Chair — Azienda Ospedaliera di Lecco
Locations (12):
- Hospital Erasme, Brussels, Belgium
- France (2):
  - Dept. of Nephrology and Dialysis Centre Pasteur Vallery Radat, Paris
  - Civil Hospital Bretagne Atlantique, Vannes
- Clinic of Internal Medicine, Rostock, Germany
- Italy (7):
  - Nephrology and Dialysis Unit Ospedali Riuniti, Ancona
  - UO Nefrologia Dialisi e Trapianto Policlinico S. Orsola Malpighi, Bologna
  - Civil Hospital, Cirié
  - PO Lastaria, Foggia
  - Hospital Maggiore della Carità, Novara
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale San Giovanni Bosco, Torino
- Hospital Val d'Hebron, Barcelona, Spain

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822